CLINICAL TRIAL: NCT01630369
Title: Multicenter, Open, Non-randomized 6 Months Study to Evaluate Efficacy and Safety Insuman® Basal, Insuman® Comb 25, Insuman® Rapid in Insulin-naÏve Patients With T2DM Who Received Baseline Education Course in the Diabetes School.
Brief Title: Efficacy and Safety of Insuman Basal/Comb/Rapid in Patients With Type 2 Diabetes
Acronym: SPIRIT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUBIN_L_05574; U1111-1128-8605 (Other: UTN)
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Human Insulin (Experimental): Dosage of human insulin (Insuman Basal/Comb/Rapid) will be individually adjusted in accordance with the Summary of Product Characteristics (SmPC). Patients will follow the titration algorithm recommended by the physician.
  Interventions: Drug: insulin human (HR1799)

INTERVENTIONS:
Drug: insulin human (HR1799) — Pharmaceutical form: solution for injection Route of administration: subcutaneous
  Other Names: Insuman Basal / Insuman Comb / Insuman Rapid

SUMMARY:
Primary Objective:

- To evaluate the decrease of Hb A1c ≥ 1% after 6 month treatment in patients with Type 2 Diabetes Mellitus (T2DM) uncontrolled on Oral Antidiabetics (OADs)

Secondary Objectives:

* To evaluate the percentage of patients with Hb A1c < 7.5%,
* To evaluate the rate of hypoglycaemia (symptomatic, severe)
* To evaluate the middle dose of insulin per product - Insuman Basal, Insuman Comb, Insuman Rapid after 6 month treatment
* To evaluate the change in Fasting Plasma Glucose (FPG) after 6 month treatment
* To assess the overall safety
* To evaluate the efficacy of education courses in Diabetes Schools (% of correct answers after second test compare to the testing of the initial level)

DETAILED DESCRIPTION:
6 months

ELIGIBILITY:
Inclusion criteria :

* T2DM patients uncontrolled by maximum tolerated dose of 1-2 OADs
* Males and Female > 18 years
* HbA1c > 7.5%
* Patients with abilities of self-monitoring of Diabetes, managing of patient's diary, ability to obtain education in Diabetes School, completion of Questionnaire
* It is expected that the patient will remain on a stable dose of OADs within 6 months of treatment

Exclusion criteria :

* Type 1 diabetes
* Current temporary insulin therapy (gestational diabetes, pancreas cancer, surgery, clinical trial)
* Any clinically significant acute major organ or systemic diseases making interpretation of the evaluation results difficult
* Patient planning a pregnancy now or in the next 6 months
* The patient is participating in another clinical study now or in the last 28 days prior to Visit 1
* The patient is a drug user (currently or in the past)

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 552 (Actual)
Dates: Start 2012-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Decrease of Hb A1c ≥ 1% | Baseline, 6 months

SECONDARY OUTCOMES:
Percentage of patients with Hb A1c < 7.5% | 6 months
Rate of hypoglycaemias (symptomatic, severe) | 6 months
Middle dose of insulin per product (Insuman Basal, Insuman Comb, Insuman Rapid) | 6 months
Change in FPG | Baseline 6 months
Number of patients with adverse events | 6 months
Assessment of efficacy of education courses in Diabetes Schools | Baseline, 6 months
  Percentage of correct answers after second test compare to the testing of the initial level

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Kyiv, Ukraine